CLINICAL TRIAL: NCT03021252
Title: The RETORNUS-2 Study: Impact of Respiratory Muscle Training on Swallowing Disorders in Stroke Patients
Brief Title: Respiratory Muscle Training in Stroke Swallowing Disorders
Acronym: RETORNUS-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the SARS-COV2 pandemic. Recruitment stopped at 48 patients
Sponsor: Parc de Salut Mar (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSM/RHB/NR21
Record Dates: First submitted 2017-01-10; First posted 2017-01-13 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2019-09

CONDITIONS: Swallowing Disorder; Stroke; Respiratory Muscle Training; Malnutrition
MeSH Terms: conditions — Deglutition Disorders; Stroke; Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity IEMT (Experimental): Inspiratory and expiratory muscle training + standard swallow therapy.
  Interventions: Device: High intensity IEMT
- Sham IEMT (Sham Comparator): Sham inspiratory and expiratory muscle training + standard swallow therapy
  Interventions: Device: Sham IEMT

INTERVENTIONS:
Device: High intensity IEMT — Training load will be the maximum inspiratory / expiratory load defined according to patient tolerance equivalent to 10 maximal repetitions (RM) as 10 consecutive inspirations / expirations (x 5 set), three times per day, during 8 weeks. External loads will be increased weekly at intervals of 10 cm H2O as tolerated. Patients will receive standard swallow therapy consisting of swallowing manoeuvres, oral exercises, and compensatory techniques aimed to improve self-management of dysphagia and protect the airway.
  Arms: High intensity IEMT
Device: Sham IEMT — 5 sets of 10 inspirations and expirations in a sham IEMT trainer, three times a day, during 8 weeks.
  Arms: Sham IEMT

SUMMARY:
Clinical randomized clinical trial to assess the effectiveness of incorporating inspiratory and expiratory muscle training (IEMT) in the rehabilitation of stroke patients with dysphagia in terms of functional outcomes, comorbidities, survival and quality of life.

This project also incorporates a longitudinal study to assess the clinical impact of dysphagia on body composition and nutritional status in stroke patients.

DETAILED DESCRIPTION:
Stroke is a major cause of morbidity and mortality worldwide. Stroke can lead to varying degrees of oropharyngeal dysphagia (25-85% of patients) and respiratory muscle dysfunction associated with an increase in medical complications such as bronchoaspiration, malnutrition and death. Dysphagia is present in a significant proportion of patients admitted to Rehabilitation (up to 85% depending on series) in stroke. Standard swallow therapy consists of educational intervention aimed to improve self-management of dysphagia and protect the airway, oral exercises to improve lingual praxis, and compensatory techniques based on videofluoroscopic findings. Recent studies suggest that IEMT can improve swallowing efficacy and reduce eventual bronchoaspiration events.

Nutritional status appears in 9-67% of patients with acute and subacute stroke and has an impact on functional outcomes and provides information about the risk of hospitalization and death. Stroke patients are at risk of developing malnutrition because of neurologic impairments related to feeding (chewing, deglutition and self-feeding) that can result in a poor food intake. To date, there is only few studies on prevalence and influence of malnutrition in stroke.

ELIGIBILITY:
Inclusion Criteria:

* First-ever Ischemic or haemorrhagic stroke
* Time since stroke onset: 1 month
* Dysphagia confirmed by videofluoroscopic study with a score >3 in the 8-point Penetration Aspiration Scale.
* Mini-mental State Exploration > 24)

Exclusion Criteria:

* Aphasia
* History of cardiopulmonary disease; neurologic condition other than stroke and metabolic disease
* Medical treatment with potential effect on muscle structure and function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Change in respiratory muscle strength | Baseline and weekly during 8 weeks
  Respiratory muscle strength is assessed through maximal inspiratory and expiratory pressures (PImax and PEmax, respectively) using a pressure transducer connected to a digital register system. The PImax is measured at mouth during a maximum effort from residual volume against occluded airway. To determine the PEmax, the patients will perform a maximum expiratory effort from total lung capacity (TLC) in the face of the occluded airway. A specific and validated respiratory pressures manometer will be used (Micro RPM, Cardinalhealth, Kent, UK).
Change in dysphagia severity | Baseline, 8 weeks, 6 months post-stroke
  Dysphagia severity is assessed with the Penetration-Aspiration Scale: scores of 1-2 indicate normal swallowing; 3-5, penetration; >6, aspiration.

SECONDARY OUTCOMES:
Change in tongue strength | Baseline and weekly during 8 weeks
  Lingual Force (IOPI system): maximum isometric tongue pressure defined as the highest of the three peak isometric tongue pressure scores.
Change in fat-free mass | Baseline, 3 months and 6 months post-stroke
  Fat-free mass measured by electrical bioimpedance in kilograms and expressed as normal, low or high values according to normal values for the reference population
Malnutrition at 6 months | Baseline and 6 months post-stroke
  Malnutrition criteria of the European Society of Clinical Nutrition and Metabolism (ESPEN)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Guillén-Solà, MD, PhD, Principal Investigator — Fundació IMIM - Parc de Salut Mar
Locations (2):
- Spain (2):
  - Hospital de l'Esperança, Barcelona, Catalonia
  - Physical Medicine & Rehabilitation Dpt. Parc de Salut Mar., Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Guillen-Sola A, Messagi Sartor M, Bofill Soler N, Duarte E, Barrera MC, Marco E. Respiratory muscle strength training and neuromuscular electrical stimulation in subacute dysphagic stroke patients: a randomized controlled trial. Clin Rehabil. 2017 Jun;31(6):761-771. doi: 10.1177/0269215516652446. Epub 2016 Jun 7. PMID 27271373
- [Background] Messaggi-Sartor M, Guillen-Sola A, Depolo M, Duarte E, Rodriguez DA, Barrera MC, Barreiro E, Escalada F, Orozco-Levi M, Marco E. Inspiratory and expiratory muscle training in subacute stroke: A randomized clinical trial. Neurology. 2015 Aug 18;85(7):564-72. doi: 10.1212/WNL.0000000000001827. Epub 2015 Jul 15. PMID 26180145
- [Background] Kulnik ST, Birring SS, Moxham J, Rafferty GF, Kalra L. Does respiratory muscle training improve cough flow in acute stroke? Pilot randomized controlled trial. Stroke. 2015 Feb;46(2):447-53. doi: 10.1161/STROKEAHA.114.007110. Epub 2014 Dec 11. PMID 25503549
- [Background] Burgos R, Sarto B, Elio I, Planas M, Forga M, Canton A, Trallero R, Munoz MJ, Perez D, Bonada A, Salo E, Lecha M, Enrich G, Salas-Salvado J; Group for the Study of Malnutrition in Hospitals in Catalonia. Prevalence of malnutrition and its etiological factors in hospitals. Nutr Hosp. 2012 Mar-Apr;27(2):469-76. doi: 10.1590/S0212-16112012000200018. PMID 22732970
- [Derived] Guillen-Sola A, Messaggi-Sartor M, Ramirez-Fuentes C, Marco E, Duarte E. The Retornus-2 study: impact of respiratory muscle training in subacute stroke patients with dysphagia, study protocol of a double-blind randomized controlled trial. Trials. 2021 Jun 25;22(1):416. doi: 10.1186/s13063-021-05353-y. PMID 34172071